CLINICAL TRIAL: NCT00056173
Title: A Phase I/II Study of GTI-2040 and Capecitabine Combination Therapy in Patients With Advanced or Metastatic Renal Cell Carcinoma (mRCC)
Brief Title: Combination of Capecitabine and GTI-2040 in the Treatment of Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aptose Biosciences Inc. (Industry)
Collaborators: Wake Forest University (Other); University of Chicago (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L01-1409; NCT00084331 (obsolete NCT alias)
Record Dates: First submitted 2003-03-06; First posted 2003-03-10 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Carcinoma, Renal Cell; Metastases, Neoplasm
Keywords: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — GTI2040

INTERVENTIONS:
Drug: GTI-2040

SUMMARY:
This phase II, 43 patient trial, will evaluate the efficacy of GTI-2040, an antisense oligonucleotide complementary to the R2 component of ribonucleotide reductase (RNR) mRNA, in combination with capecitabine, in the setting of advanced/metastatic renal cell carcinoma. Preclinical studies have shown synergy between GTI-2040 and capecitabine against renal cell carcinoma.

ELIGIBILITY:
* Age greater than or equal to 18.
* Histologically or cytologically confirmed diagnosis of advanced or metastatic renal cell carcinoma for which no effective therapy is available or that is unresponsive to conventional therapy.
* Measurable disease. To be considered measurable, a lesion must be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral CT scan.
* Karnofsky performance status of greater than or equal to 70.
* Be able to have a central venous like access maintained throughout the study.
* Provide written informed consent prior to the initiation of protocol therapy.
* Appropriate organ function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2002-03; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Bay Area Cancer Research Group, Concord, California
  - USC-Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - CA Hematology Oncology Medical Group, Torrance, California
  - Innovative Medical Research of South Florida, Inc., Miami Shores, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - SUNY Upstate Medical University, Syracuse, New York
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: Lorus Therapeutics Website — http://www.lorusthera.com